CLINICAL TRIAL: NCT02111369
Title: Propranolol and Botulinum Toxin for Essential Vocal Tremor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael M Johns MD, Director, Emory Voice Center, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00072929
Record Dates: First submitted 2014-04-08; First posted 2014-04-11 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Essential Vocal Tremor; Essential Voice Tremor; Essential Tremor; Voice Tremor; Vocal Tremor
Keywords: Essential Tremor; Essential Vocal Tremor; Essential Voice Tremor
MeSH Terms: conditions — Essential Tremor | interventions — Propranolol; Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propranolol/Botulinum (Experimental): After baseline analysis, patient will be given a prescription by the principal investigator for propranolol. This prescription will consist of a starting dose of generic immediate-release at 10 mg three times per day (30 mg each day) with an increase in dose in 5-7 days if there is no effect (60 mg each day) and if the patient had demonstrated no side effects. Dose may be increased to 240 mg each day depending on patient improvement and side effect profile. After second evaluation, patient will receive botulinum toxin injections. The risks and benefits of botulinum toxin therapy will be explained to the patient, and bilateral injections will take place.
  Interventions: Drug: Propranolol; Procedure: Botulinum Toxin

INTERVENTIONS:
Drug: Propranolol — After a discussion of the risks and benefits of propranolol therapy, the patient will then be given a prescription by the principal investigator for propranolol. This prescription will consist of a starting dose of generic immediate-release at 10 mg three times daily (30 mg each day) with an increase in dose in 5-7 days if there is no effect (60 mg each day) and if the patient had demonstrated no side effects. Dose may be increased to 240 mg each day depending on patient improvement and side effect profile.
  Other Names: Inderal
Procedure: Botulinum Toxin — At the second evaluation, patient will receive botulinum toxin injections. The risks and benefits of botulinum toxin therapy will be explained to the patient, and bilateral injections will take place.

SUMMARY:
Essential tremor is the most common adult-onset movement disorder, and essential voice tremor is the vocal manifestation of essential tremor. While nearly all essential tremor patients experience hand tremor, many also manifest head tremor and voice tremor. Essential voice tremor can lead to increased vocal effort, decreased intelligibility, and misconstrued emotional state. Only one medication, propranolol, is FDA-approved to treat essential tremor. Propranolol is not felt to be nearly as effective for axial tremors (head, trunk, neck) as it is for extremity tremors. However, this has not been studied with any objective assessment in a prospective way for EVT. For patients with essential voice tremor, the limited published data suggests that botulinum toxin has been shown to lead to functional voice improvement. Botulinum toxin, though also not well-studied with objective voice outcomes, is a commonly used clinical therapy for treatment of essential voice tremor. While it is used more often for essential voice tremor than propranolol therapy, botulinum toxin also has not been prospectively studied with validated, objective voice outcome measures. The investigators would like to determine if propranolol has any significant effect on vocal tremor. The investigators would also like to determine, in an objective way, the effect of botulinum toxin on vocal tremor. If effective, propranolol would provide an affordable and non-invasive alternative or addition to botulinum toxin injections for patients with essential voice tremor.

DETAILED DESCRIPTION:
Specific Aims

• Determine the effect of propranolol on vocal tremor in the treatment-seeking population.

To date, the nonselective beta-blocker propranolol remains the only agent approved for the treatment of essential tremor (ET). For ET, immediate and sustained release formations of propranolol are equally effective, while other beta-blockers like nadolol and timolol are not as effective. While propranolol improves tremor in greater than half of patients with essential tremor, its effects on tremor are not evenly distributed. Improvement in tremor symptoms is greater for limb tremor than axial tremor, and therefore propranolol is not commonly used for the treatment of essential voice tremor (EVT). However, its effect on essential voice tremor has never been objectively, prospectively studied. Our aim is to objectively determine the effect of propranolol on essential voice tremor in the treatment-seeking population by evaluating patients with EVT before and after propranolol therapy.

• Determine the effect of botulinum toxin injections on vocal tremor in the treatment-seeking population.

More recently, botulinum toxin A has been used for the treatment of EVT. Chemical denervation with botulinum toxin is only modestly effective in reducing limb tremor in ET and complicated by side effects of weakness. However, botulinum toxin seems to be more effective in treating EVT than other manifestations of ET. While prior studies have not enlisted validated assessments of voice quality to measure the effect of botulinum toxin injections on EVT, they have shown subjective improvement in acoustic measures of tremor and ratings of videotaped speech after therapy with botulinum toxin. Our aim is to objectively determine the effect of botulinum toxin on vocal tremor in the treatment-seeking population by evaluating patients with EVT before and after botulinum therapy.

Voice Evaluations and Medications

For the first evaluation, a research coordinator will collect demographics and patient reported data. This data will result from providing patient questionnaires and recording the patient's voice. VRQOL data will be collected by having the patient answer ten statements on a 1-5 scale, such as "I have trouble speaking loudly or being heard in noisy situations" or "I run out of air and need to take frequent breaths." QUEST data will be also recorded to a 30-item essential tremor-specific questionnaire. Patient will also complete a global voice rating of a 0-7 scoring of "How would you rate your voice today?" After these subjective questionnaires, patient will participate in a vocal recording using prompts and passages from the validated CAPE-V voice assessment tool.

After a discussion of the risks and benefits of propranolol therapy, the patient will then be given a prescription by the principal investigator for propranolol.

The second evaluation will occur at an office visit two weeks after initiating propranolol therapy. Again, this will consist of patient-reported V-RQOL, QUEST, and global voice rating data. Patient will participate in a second vocal recording using prompts and passages from the validated CAPE-V voice assessment tool.

At this second evaluation, patient will receive botulinum toxin injections. The risks and benefits of botulinum toxin therapy will be explained to the patient, and bilateral injections will take place.

Four weeks after botulinum toxin injection, the patient will undergo the third voice assessment. Again, this will consist of patient-reported V-RQOL, QUEST, and global voice rating data. Patient will participate in a third vocal recording using prompts and passages from the validated CAPE-V voice assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of essential voice tremor
* Patients who have received or are planning to receive botulinum toxin injections for essential voice tremor
* Patients who give informed consent to be contacted for research

Exclusion Criteria:

* Patients who are already on a beta blocker
* Patients who suffer from hypotension, bradycardia, or otherwise have a medical contraindication to beta blocker therapy (eg. moderate to severe bronchial asthma)

If the patient has received botulinum toxin injections for EVT previously, a three-month washout period is necessary before participation.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Johns, MD, Principal Investigator — Emory Voice Center
Locations (1):
- Emory Voice Center, Atlanta, Georgia, United States

REFERENCES:
- [Background] Sulica L, Louis ED. Clinical characteristics of essential voice tremor: a study of 34 cases. Laryngoscope. 2010 Mar;120(3):516-28. doi: 10.1002/lary.20702. PMID 20066728
- [Background] Zesiewicz TA, Shaw JD, Allison KG, Staffetti JS, Okun MS, Sullivan KL. Update on treatment of essential tremor. Curr Treat Options Neurol. 2013 Aug;15(4):410-23. doi: 10.1007/s11940-013-0239-4. PMID 23881742
- [Background] Gurey LE, Sinclair CF, Blitzer A. A new paradigm for the management of essential vocal tremor with botulinum toxin. Laryngoscope. 2013 Oct;123(10):2497-501. doi: 10.1002/lary.24073. Epub 2013 Apr 1. PMID 23553653
- [Background] Adler CH, Bansberg SF, Hentz JG, Ramig LO, Buder EH, Witt K, Edwards BW, Krein-Jones K, Caviness JN. Botulinum toxin type A for treating voice tremor. Arch Neurol. 2004 Sep;61(9):1416-20. doi: 10.1001/archneur.61.9.1416. PMID 15364688
- [Background] Hogikyan ND, Sethuraman G. Validation of an instrument to measure voice-related quality of life (V-RQOL). J Voice. 1999 Dec;13(4):557-69. doi: 10.1016/s0892-1997(99)80010-1. PMID 10622521
- [Background] Troster AI, Pahwa R, Fields JA, Tanner CM, Lyons KE. Quality of life in Essential Tremor Questionnaire (QUEST): development and initial validation. Parkinsonism Relat Disord. 2005 Sep;11(6):367-73. doi: 10.1016/j.parkreldis.2005.05.009. PMID 16103000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Voice Center from August 2014 to February 2015.
Pre-assignment Details: Participants who previously received botulinum toxin injections for essential voice tremor (EVT) underwent a three month washout period prior to participation.
Groups:
- Propranolol/Botulinum: After baseline analysis, patient will be given a prescription by the principal investigator for propranolol. This prescription will consist of a starting dose of generic immediate-release at 10 mg three times per day (30 mg each day) with an increase in dose in 5-7 days if there is no effect (60 mg each day) and if the patient had demonstrated no side effects. Dose may be increased to 240 mg each day depending on patient improvement and side effect profile. After second evaluation, patient will receive botulinum toxin injections. The risks and benefits of botulinum toxin therapy will be explained to the patient, and bilateral injections will take place.
  Propranolol: After a discussion of the risks and benefits of propranolol therapy, the patient will then be given a prescription by the principal investigator for propranolol. This prescription will consist of a starting dose of generic immediate-release at 10 mg three times daily (30 mg each day) with an increase in dose in 5-7 days
Period: Overall Study
Arm/Group | Propranolol/Botulinum
Started | 18
Completed | 15
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Propranolol/Botulinum: After baseline analysis, participants were given a prescription by the principal investigator for propranolol. This prescription consisted of a starting dose of generic immediate-release at 10 mg three times per day (30 mg each day) with an increase in dose in 5-7 days if there is no effect (60 mg each day) and if the participant demonstrated no side effects. Dose was increased up to 240 mg a day depending on participant improvement and side effect profile. After second evaluation, participants received botulinum toxin injections. The risks and benefits of botulinum toxin therapy were explained to the participant, and bilateral injections took place.
Arm/Group | Propranolol/Botulinum
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life in Essential Tremor (QUEST) Questionnaire Score
Description: The QUEST questionnaire is a 30 item self-reported essential tremor-specific quality of life scale that asks participants to rate responses (never/no, rarely, sometimes, frequently, always/yes, or not applicable). Total scores range between 0 to 100 where 0 is the best score and 100 is the worst score. A higher score indicates a lower quality of life.
Time Frame: Baseline, 2 weeks, 6 weeks
Population: Participants who completed all three study visits (Baseline Visit 1, Visit 2, and Visit 3).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Propranolol/Botulinum: After baseline analysis, participants were given a prescription by the principal investigator for propranolol. This prescription consisted of a starting dose of generic immediate-release at 10 mg three times per day (30 mg each day) with an increase in dose in 5-7 days if there is no effect (60 mg each day) and if the participant demonstrated no side effects. Dose was increased up to 240 mg a day depending on participant improvement and side effect profile. After second evaluation, participants received botulinum toxin injections. The risks and benefits of botulinum toxin therapy were explained to the participant, and bilateral injections took place.
  Propranolol: After a discussion of the risks and benefits of propranolol therapy, the patient will then be given a prescription by the principal investigator for propranolol. This prescription will consist of a starting dose of generic immediate-release at 10 mg three times daily (30 mg each day) with an increase in dose in 5-7 days
Arm/Group | Propranolol/Botulinum
Number analyzed (Participants) | 15
units on a scale
  Baseline (Visit 1) | 39.41 (27.89)
  Visit 2 | 29.50 (23.73)
  Visit 3 | 23.60 (24.49)

2. Primary Outcome: Change in Voice-Related Quality Of Life (VRQOL) Questionnaire Score
Description: The VRQOL is a ten question self-reported measure that asks patients to rate responses from 1-5 (1=none, not a problem, 2=a small amount, 3=a moderate (medium) amount, 4=a lot, 5=problem is as "bad as it can be"). Total scores range from 0 to 100. A higher score indicates more problems interfering with day to day activities.
Time Frame: Baseline, 2 weeks, 6 weeks
Population: Participants who completed all three study visits (Baseline Visit 1, Visit 2, and Visit 3).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol/Botulinum
Number analyzed (Participants) | 15
units on a scale
  Baseline (Visit 1) | 42.22 (23.64)
  Visit 2 | 51.53 (26.21)
  Visit 3 | 64.16 (22.23)

3. Primary Outcome: Change in Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) Score
Description: The CAPE-V is a clinically validated perceptual voice assessment tool that is used to describe the severity of auditory-perceptual attributes of a voice problem, in a way that can be communicated among clinicians. Participant's speech is recorded and evaluated by trained "listeners". Listeners indicate overall tremor severity by making a tick mark on a 1 to 100 mm visual analog scale. Total scores range from 0 to 100 where 0 is the best score and 100 is the worst score.
Time Frame: Baseline, 2 weeks, 6 weeks
Population: Participants who completed all three study visits (Baseline Visit 1, Visit 2, and Visit 3).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol/Botulinum
Number analyzed (Participants) | 15
units on a scale
  Baseline (Visit 1) | 43.61 (23.26)
  Visit 2 | 45.89 (24.57)
  Visit 3 | 35.67 (22.14)

4. Primary Outcome: Change in Global Voice Rating
Description: Patient-Reported Measure
  • 0-7 ranking
Time Frame: Baseline, 2 weeks, 6 weeks
Population: Data were not collected as investigators found the Voice Related Quality of Life (VRQOL) scale to be a better measure.
Arm/Group | Propranolol/Botulinum
Number analyzed (Participants) | 0

5. Primary Outcome: Change in Acoustic Spectrograms
Description: Objective Voice Assessment
  • Using the Computerized Speech Laboratory speech and voice analysis system (KayPENTAX, Montvale, NJ)
Time Frame: baseline, 2 weeks, 6 weeks
Population: Data were not collected as investigators found the Voice Related Quality of Life (VRQOL) scale to be a better measure.
Arm/Group | Propranolol/Botulinum
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Propranolol/Botulinum
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
The study lacks a placebo or control group, with participants representing their own internal controls. Additionally, inter-rater reliability among listeners for the CAPE-V outcome measure analysis was low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No